CLINICAL TRIAL: NCT00368615
Title: Characterization of the Melanoma-Specific Immune Response
Acronym: Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 362163
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Melanoma
Keywords: melanoma; malignant melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood will be collected prior to initiation of chemotherapy. There will be no more than two blood draws per subject. Most subjects will receive a single blood draw; however, some may be asked to return for an additional blood draw if investigators were unable to isolate melanoma-specific immune cells after the first blood draw. Two separate blood draws will be the maximum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects ages 18-85 years old with biopsy proven melanoma. Peripheral blood will be collected from adults ages 18-85 years old. These samples will then be used for PCR analysis and to generate melanoma-specific T cell clones. If the participant requires a palliative resection of a melanoma tumor(s) then tissue from the tumor will be used to characterize the melanoma's interaction with the immune system and to generate melanoma-specific cell lines. T cell clones isolated from participant's peripheral blood will then be assayed for in-vitro responsiveness to these cell lines. All experiments will be conducted in-vitro.
- 2: Age-matched controls (no evidence of melanoma)

SUMMARY:
The aim of this study is to study T-cells. Blood will be collected and the samples will be used to generate T cell clones. Two separate blood draws will be required at the maximum.

DETAILED DESCRIPTION:
The aim of the study is to in-vitro characterize and expand T cells specific for melanoma-derived antigens. Peripheral blood with be collected from 20 volunteers with biopsy proven melanoma and 10 age matched controls. Blood will be collected prior to the initiation of chemotherapy. There will be no more than two blood draws per patient. Most patients will receive a single blood draw; however, some participants may be asked to return for a single additional blood draw if investigators were unable to isolate melanoma-specific immune cells after the first blood draw. Two separate blood draws will be the maximum. The interval between these blood draws will be a minimum of 3 months apart. Blood samples will be used to determine the patient's HLA haplotype via PCR and DNA sequencing. After the patient's haplotype has been established melanoma-specific T cell clones will be generated from the peripheral blood samples and expanded in-vitro. These clones will then be assayed for specificity against commercially available melanoma cell lines. The T cell clones will also be assayed for reactivity to melanocyte differentiation antigens such as MART-1 and gp100. If the volunteer requires a palliative resection of a melanoma tumor then the patient's own tumor cells may also be used to test the specificity of the isolated T cell clones. All experiments will be conducted in-vitro.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy diagnosis of malignant melanoma
* Have had a biopsy diagnosis of malignant melanoma in the past

Exclusion Criteria:

* Patients taking immunosuppressive medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 years to 85 years who have a biopsy diagnosis of melanoma, and age-matched controls (subjects who do not have a diagnosis of melanoma).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-08; Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
melanoma - peripheral blood | 2 Years
  Peripheral blood will be collected from adults ages 18-85 years old. These samples will then be used for PCR analysis and to generate melanoma-specific T cell clones. If the participant requires a palliative resection of a melanoma tumor(s) then tissue from the tumor will be used to characterize the melanoma's interaction with the immune system and to generate melanoma-specific cell lines. T cell clones isolated from participant's peripheral blood will then be assayed for in-vitro responsiveness to these cell lines. All experiments will be conducted in-vitro.

SECONDARY OUTCOMES:
melanoma - biopsy | 2 Years
  Patients will not be required to have a biopsy to participate in the study but those who give their consent will undergo a skin biopsy. The biopsy will be used to characterize the skin-infiltrating inflammatory cells. The gene-expression profile of these cells will be determined. Each patient who provides consent will undergo two biopsies, one of lesional skin and the other of normal lesional skin as control. Patients who develop multiple cutaneous tumors may be reconsented for an additional two biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical
- See also: Learn more or sign up for the study here! — https://studypages.com/s/determining-how-melanoma-interacts-with-the-immune-system-999173/